CLINICAL TRIAL: NCT02253667
Title: Palliative Use of High-flow Oxygen Nasal Cannula in End-of-life Patients: a Randomized Controlled Trial
Brief Title: Palliative Use of High-flow Oxygen Nasal Cannula in End-of-life Lung Disease Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: One of the investigators left the department, Master Degree in which this study was part of her thesis. No patients were enrolled.
Sponsor: Hospital Sao Joao (Other)
Responsible Party: Principal Investigator, Miguel R. Goncalves, Clinical Professor, PH.D, Hospital Sao Joao
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PalliativeHFONC
Record Dates: First submitted 2014-09-28; First posted 2014-10-01 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Lung Disease; Acute Respiratory Distress Syndrome
Keywords: Palliative care; Lung disease; Acute Respiratory Distress Syndrome; High-flow oxygen nasal cannula; Dyspnoea; Opioids
MeSH Terms: conditions — Lung Diseases; Respiratory Distress Syndrome; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HFONC (Experimental): Patient will use HFONC with FiO2 enough to achieve SpO2>90%. If needed, morphine is titrated to reduce a patient's dyspnoea score by at least one point on the Borg scale and to achieve at least level 5 or less. Initial dose: 10 mg, repeated every 4h until the desired reduction in dyspnoea is obtained. In the case of refractory dyspnoea, the dose is increased by 50%.
  Interventions: Device: HFONC
- Conventional oxygen (Other): Patient will use venturi or reservoir mask with FiO2 enough to achieve SpO2>90%. If needed, morphine is titrated to reduce a patient's dyspnoea score by at least one point on the Borg scale and to achieve at least level 5 or less. Initial dose: 10 mg, repeated every 4h until the desired reduction in dyspnoea is obtained. In the case of refractory dyspnoea, the dose is increased by 50%.
  Interventions: Device: Conventional oxygen therapy

INTERVENTIONS:
Device: HFONC
  Other Names: Optiflow (Fisher&Paykel ™)
  Arms: HFONC
Device: Conventional oxygen therapy
  Other Names: Venturi mask; Reservoir mask
  Arms: Conventional oxygen

SUMMARY:
The prevalence of severe dyspnoea among terminally ill patients has been reported as 70% and 90% for lung cancer and chronic obstructive pulmonary disease (COPD) patients, respectively.

Current management to dyspnoea includes opioids, psychotropic drugs, inhaled frusemide, Heliox 28 and oxygen.

Conventional oxygen supplementation is often used in these patients, but it may be inadequate, especially if they require high flows (from 30L/min to 120L/min in acute respiratory failure).

High-flow oxygen nasal cannula (HFONC) is a new technological device in high-flow oxygen system that consists of an air-oxygen blender (allowing from 21% to 100% FiO2) which generates the gas flow rate up to 55 L/min and a heated humidification system. This technology may have an important role in reducing respiratory distress in do-not-intubate patients.

Some HFONC's beneficial effects are the washout of the nasopharyngeal dead space reducing rebreathing of CO2 and improvement oxygenation through greater alveolar oxygen concentration; a better matching between patient's inspiratory demand and oxygen flow; generation of a certain level of positive pressure (PEEP) contributing to the pulmonary distending pressure and recruitment; improvement of lung and airway mucociliary clearance due to the heated and humidified oxygen; and patient's comfort because of the nasal interface allowing feeding and speech.

The investigators hypothesize that patients supported with HFONC need less opioids to decrease dyspnoea.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients who had end-stage lung disease (lung cancer, pulmonary fibrosis, COPD, …) - (McCabe score > 3 [<6 months life expectancy] and a Palliative Prognostic Index score ≥ 4) admitted to hospital because of acute respiratory failure and distress
* Had chosen to forego all life support and receiving only palliative care
* Severe hypoxemia (PaO2/FiO2< 250)
* At least one of the following: dyspnoea (Borg scale ≥4), signs of respiratory distress, and respiratory rate greater than 30 beats per min

Exclusion Criteria:

* Patients had to be competent (Kelly score <4)
* Refusal of treatment
* Weak cough reflex
* Agitation or non-cooperation
* Uncontrolled cardiac ischemia or arrhythmias
* Failure of more than two organs
* Use of opioids within the past 2 weeks
* Adverse reactions to opioids
* History of substance misuse
* Known contraindication for morphine (acute renal failure and recent head injury)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Dyspnoea | 2 days
  We aim to reduce dyspnoea more effective, using Borg Scale, with HFONC compared to conventional oxygen mask.
Opioids | 2 days
  By randomizing the two groups we will be able to compare the total use of opioids.

SECONDARY OUTCOMES:
Physiologic variables | 2 days
  The comparison in respiratory rate, heart rate, mean arterial pressure and oxygen saturation between the two groups.
Patient comfort | 2 days
  Detect if there is a difference in patient comfort using HFONC or conventional oxygen mask.
Mortality | 6 months
  Overall mortality in hospital and at 3 months and 6 months after discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel R Gonçalves, PhD, Principal Investigator — Pulmonology Department, University Hospital São João
Locations (1):
- University Hospital of São João, Porto, Porto District, Portugal